CLINICAL TRIAL: NCT04056702
Title: Impact of Elexacaftor-tezacaftor-ivacaftor Triple Combination CFTR Therapy on Sinus Disease: Quantitative Sinus Computed Tomography, Patient Reported Outcomes and Cellular and Molecular Changes
Brief Title: Impact of Triple Combination CFTR Therapy on Sinus Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jennifer Taylor-Cousar (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Jennifer Taylor-Cousar, Professor of Medicine, National Jewish Health
Organization: National Jewish Health (Other)
Other Study IDs: HS-3236
Record Dates: First submitted 2019-07-27; First posted 2019-08-14 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis
Keywords: Chronic Sinusitis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Prescribed triple combination: A group of 60 people with CF who are clinically prescribed elexacaftor-tezacaftor-ivacaftor and have chronic sinusitis
  Interventions: Drug: Elexacaftor-tezacaftor-ivacaftor exposure
- Not eligible for modulators: A group of 10 patients with two class I/II mutations who are ineligible for elexacaftor-tezacaftor-ivacaftor based on their genotype and have chronic sinusitis.

INTERVENTIONS:
Drug: Elexacaftor-tezacaftor-ivacaftor exposure — Once a clinical decision has been made to prescribed a patient triple combination therapy, people with CF are eligible to participate in this study.
  Groups: Prescribed triple combination

SUMMARY:
The study's main goal is to observe how effective elexacaftor-tezacaftor-ivacaftor is for improving the symptoms and signs of CF-related sinus disease.

DETAILED DESCRIPTION:
To determine if elexacfator-tezacaftor-ivacaftor improves the signs and symptoms of CF-related sinus disease, before and after initiation of triple combination therapy, each subject will undergo sinus CT scan and complete questionnaires related to signs and symptoms of sinus disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects from 18 to 89 years old.
2. Subjects with cystic fibrosis and comorbid chronic sinus disease (historic diagnosis based on physician assessment of signs and symptoms and medical record).
3. Subjects who clinically elect to initiate elexacaftor-tezacaftor-ivacaftor therapy and/or that are ineligible for CFTR modulator therapy based on their genotype, but have class I/II mutations based on sweat chloride > 90 mmol/L.

Exclusion Criteria:

1. Subjects under the age of 18 or over the age of 89.
2. Subjects who do not elect to initiate elexacaftor-tezacaftor-ivacaftor for clinical reasons.
3. Subjects who had sinus surgery within the last 6 months or will have sinus surgery during the study period.
4. Subjects who have had a recent pulmonary exacerbation or viral infection within two weeks of initial visit.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with cystic fibrosis and chronic sinusitis.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in Sinus CT opacification. | Change in Sinus CT opacification between the initial and 6 month visits.
  Calculated from an automated quantification of the size of sinuses.

SECONDARY OUTCOMES:
Change in 22-item Sino-Nasal Outcome Test (SNOT-22) score. | Change in SNOT-22 score between the initial and 6 month visits.
  Validated, disease-specific measure of sinus symptoms. Contains 22 questions that are all scored from 0 to 5, when summed a total score ranges form 0 to 110. Higher scores represent worse sinus symptoms.
Change in Questionnaire for Olfactory Disorders (QOD) score | Change in QOD score between the initial and 6 month visits.
  Validated, disease-specific measure of olfaction, i.e. the ability to smell. Contains 19 questions that are scored form 0 to 3, when summed a total score can range form 0 to 57. Higher scores indicate greater impact on a subjects sense of smell.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer TaylorCousar, M.D., Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No